CLINICAL TRIAL: NCT07267988
Title: Additional Effects Of Brandt-Daroff Exercises With GANS Maneuver On Dizziness And Quality Of Life In Patients With BPPV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/12
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: BPPV; Dizziness; Quality of Life
Keywords: Dizziness; BPPV; Postural pain; Quality of life
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GANS Maneuver with Brand-Daroff Exercises (Experimental): GANS Maneuver include:
  1. Sit upright on a bed with legs extended.
  2. Turn patient head 45° toward the affected ear.
  3. Quickly lie back so patient head is slightly hanging over the edge
  4. Hold this position 30-60 seconds or until vertigo stops.
  5. Without lifting the head, rotate it 90° toward the opposite side (45° past midline).
  6. Hold again for 30-60 seconds.
  7. Continue turning patient head in the same direction and roll onto side so nose faces the floor.
  8. Hold 30-60 seconds.
  9. Sit up slowly, keeping patient chin slightly tucked.
  10. Rest in sitting for about a minute. (3 reps/2 times per week) BRANDTDAROFF EXERCISES Sit upright on the edge of your bed. Turn your head 45° to the left. Keeping the head turned, quickly lie down on your right side. Hold this position 30 seconds or until vertigo stops. Return to sitting; hold 30 seconds. Turn your head 45° to the right. Quickly lie down on your left side. Hold 30 seconds or until vertigo stops. Return to sitting; hold 30 seconds.
  Interventions: Procedure: GANS Maneuver with Brandt-Daroff Exercises
- GANS Maneuver (Active Comparator): GANS Maneuver include:
  1. Sit upright on a bed with legs extended.
  2. Turn patient head 45° toward the affected ear.
  3. Quickly lie back so patient head is slightly hanging over the edge
  4. Hold this position 30-60 seconds or until vertigo stops.
  5. Without lifting the head, rotate it 90° toward the opposite side (45° past midline).
  6. Hold again for 30-60 seconds.
  7. Continue turning patient head in the same direction and roll onto side so nose faces the floor.
  8. Hold 30-60 seconds.
  9. Sit up slowly, keeping patient chin slightly tucked.
  10. Rest in sitting for about a minute. (3 reps/2 times per week)
  Interventions: Procedure: Gans Maneuver

INTERVENTIONS:
Procedure: GANS Maneuver with Brandt-Daroff Exercises — The intervention program spans six weeks and involves both supervised Gans Maneuver sessions and home-based Brandt-Daroff exercises. Participants will attend two supervised Gans sessions per week, with each session consisting of three repetitions of the maneuver.
  In addition, participants will perform Brandt-Daroff exercises at home twice daily, with each cycle consisting of three repetitions. This combination of supervised and home-based practice will be maintained consistently throughout all six weeks. Across the entire program, participants will complete a total of 12 supervised Gans sessions and 36 Brandt-Daroff home sessions.
  Arms: GANS Maneuver with Brand-Daroff Exercises
Procedure: Gans Maneuver — The control group will participate in a structured six-week intervention program consisting exclusively of the Gans Maneuver. Participants will attend two supervised sessions per week, ensuring consistent oversight and proper technique throughout the program. Each session will include three repetitions of the maneuver, with participants allowed a rest period of 30 to 60 seconds between repetitions to prevent fatigue and maintain the quality of each movement. This frequency and volume are maintained consistently across all six weeks to provide a standardized exposure, allowing for accurate comparison with other intervention groups. Over the entire six-week period, participants will complete a total of 12 supervised sessions, each with three repetitions, summing up to 36 repetitions across the intervention.
  Arms: GANS Maneuver

SUMMARY:
Benign Paroxysmal Positional Vertigo (BPPV) is the most common cause of recurrent vertigo, with a lifetime prevalence of about 2.4% and a yearly incidence of roughly 0.6%. It results from displaced otoconia within the semicircular canals and is especially common in older adults. BPPV leads to brief, position-provoked episodes of vertigo, dizziness, and imbalance, and reduced quality of life. Although canalith-repositioning maneuvers are highly effective, recurrence is common, emphasizing the need for supportive and adjunctive management strategies.This randomized controlled trial will evaluate the Additional Effects OF Brandt-Daroff Exercise With GANS Maneuver On dizziness And Quality of Life In Patients with BPPV. Thirty patients with BPPV will be recruited at Fauji Foundation Hospital and screened using the Dizziness Handicap Inverntory Scale(DHI) and Vestibular Activities and Participation measure(VAP). Participants will be randomized into two groups: (1) Reciving GANS Manuever Alone (2) GANS Manuever with Brandt-Daroff Exercises(3 sessions per week/40minutes). Dizziness will be assessed using the Dizziness Handicap Inverntory Scale(DHI) , quality of life using the Activities and Participation Measure(VAP) Scale. Outcome measures will be recorded at baseline and post-intervention. Ethical approval will be obtained from FUMC ERC, and data will be analyzed using SPSS v.22.

DETAILED DESCRIPTION:
Benign Paroxysmal Positional Vertigo (BPPV) is a common and disabling vestibular disorder, affecting approximately 2.4% of individuals during their lifetime and accounting for nearly 20-30% of vertigo cases in clinical settings. It is caused by the displacement of otoconia into the semicircular canals, leading to brief episodes of vertigo and dizziness, that significantly disrupt daily activities and reduce quality of life. The high prevalence of BPPV is associated with increased risks of falls, functional limitations, and recurrent episodes. Although canalith repositioning maneuvers serve as the primary treatment, recurrence rates remain substantial, underscoring the need for adjunctive therapeutic approaches that address persistent vertigo and improve overall functional outcomes.This study aims to investigate the additional effects GANS maneuver and Brandt-Daroff exercise on dizziness reduction, and quality of life improvement, in BPPV Patients .A randomized controlled trial will be conducted with participants diagnosed with BPPV.This study will be a non blinded, randomized controlled trial with two groups: the intervention group, which will receive GANS Maneuver with Brandt-Daroff Exercises, and the control group, which will receive GANS Maneuver alone. The intervention will last for six weeks, with participants attending two 40-minute sessions per week. A total of 30 individuals with BPPV will be recruited and randomly assigned to one of the two groups. The Dizziness Handicap Inventory Scale(DHI) will be used to screen for dizziness. Quality of life will be measured using the Vestibular and Participation Scale(VAP).The study will be conducted over a period of 1 year at Fauji Foundation Hospital. Ethical approval will be obtained from FUMC ERC. Recruited participants will be allocated to either group through a random sampling method. Outcome measurements will be taken at baseline and again after the 6-week intervention period. Individuals meeting the inclusion criteria will be selected, and written informed consent will be obtained after explaining the study's purpose. Data will be entered and analyzed on SPSS v. 22.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Patients of Benign Paroxysmal Vertigo (BPPV)
* Age between 18-60
* Acute and Chronic BPPV Patients
* Positive Dix-Hallpike Test
* DHI Scale: Mild-Severe (0-100)

Exclusion Criteria:

* Patients with a history of vestibular surgery or cochlear
* Patients with a history of seizures or epilepsy
* Patients with a pacemaker or implantable cardioverter-defibrillator (ICD)
* Patients with a history of severe head injury or concussion within the past year
* No other vestibular disorders or conditions that may affect balance (e.g., Meniere's disease, labyrinthitis
* No musculoskeletal or neurological conditions that may affect balance (e.g., stroke, Parkinson's disease)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Dizziness | 6 weeks
  Dizziness Handicap Inventory Scale(DHI): 25 Items (scoring16-54) where 16-34 = Mild handicap , 36-52 = moderate handicap , 52+ = severe handicap
Quality Of Life In BPPV patients | 6 weeks
  Vestibular Activities and Participation Scale (VAP): A 34-item, (1-4 score) , 1 = mild limitations, 2 = moderate limitation, and 3 = severe limitations, 4=extreme limitation

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan